CLINICAL TRIAL: NCT03989921
Title: Ovarian Reserve and Embryo Implantation
Acronym: IRO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2018/OP-01
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Ovarian Reserve; IVF

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normo responders: that have an AMH dosage greater than or equal to 1.2 ng/mL
  Interventions: Other: no intervention. observational study
- poor responders: with a dosage of less than 1.2 ng/mL
  Interventions: Other: no intervention. observational study

INTERVENTIONS:
Other: no intervention. observational study — no intervention. observational study

SUMMARY:
Compare, in young patients with In vitro fertilization (IVF), the rate of embryo implantation by early culture transfer (J2-J3) between 2 groups of patients: "normo responders" vs. "poor responders".

ELIGIBILITY:
Inclusion Criteria:

* IVF patient managed with or without ICSI between 01/01/2014 and 30/06/2015 in one of the two study centres
* Age < 35 years old
* Fresh transfer of at least one embryo between D2 and D6
* patients who have already received one or more transfer attempts.

Exclusion Criteria:

* No fresh transfer (Freeze All, segmentation failure, stimulation failure)
* Double successive embryo transfer (e. g. J3-J5). We did not retain these cases because if only one of the 2 embryos is implanted, it is not possible to know which transfer it corresponds to.
* Maternal serum FSH determination < 4 IU/ml at D3 in the baseline balance sheet (hypogonadotropic hypogonadism)

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population concerned is all young patients, defined as being under 35 years old, who have benefited from IVF in the 2 inclusion centres (Centres d'Aide Médicale à la Procréation des CHU de Nîmes and the Saint Roch clinic in Montpellier) between 01/01/2014 and 30/06/2015.
Sampling Method: Non-Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
The embryo implantation rate at 5 weeks after transfer is defined by the presence of an embryo with objective cardiac activity by ultrasound | 5weeks
  The embryo implantation rate corresponds to the number of embryos with cardiac activity found on the number of embryos transferred

CONTACTS AND LOCATIONS:
Locations (1):
- CHUNimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: Undecided